CLINICAL TRIAL: NCT03770390
Title: Cardiorespiratory Assessment and Quality of Life After Surgical Correction of Congenital Wall Malformations
Acronym: HeartSoar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL18_0184; 2018-A01574-51 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2018-12-04; First posted 2018-12-10 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Funnel Chest
MeSH Terms: conditions — Funnel Chest

STUDY DESIGN:
Intervention Model Description: This single group study documents changes before and after surgical correction of pectus excavatum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- The study population (Other): Patients included in this study have pectus excavatum. The have either already undergone corrective surgery during the four years prior to the inclusion period, or are scheduled for surgery during the inclusion period.
  Intervention: Surgical correction of pectus excavatum
  Interventions: Procedure: Surgical correction of pectus excavatum

INTERVENTIONS:
Procedure: Surgical correction of pectus excavatum — Surgical correction of pectus excavatum

SUMMARY:
The main objective of this study is to characterize the cardiorespiratory functional gain in patients with pectus excavatum following corrective surgery.

DETAILED DESCRIPTION:
The secondary objectives are:

* To measure the quality of life of patients operated on for pectus excavatum
* Identify and describe post-operative complications
* Follow-up on the body mass index changes post-surgery
* Evaluate intraoperative hemodynamic parameters before and after the retrosternal bar is placed non-invasively

ELIGIBILITY:
Inclusion Criteria:

* Patient with pectus excavatum
* The patient received corrective surgery within four years of enrollment and is scheduled for a follow-up visit --OR-- the patient is scheduled for corrective surgery during the inclusion period
* Collection of informed written consent (patient and legal guardian, if applicable)
* Obligation of affiliation or beneficiary of a social security programme

Exclusion Criteria:

* Impossibility for the patient to participate in his/her next annual follow-up visit
* Absence of exercise test data AND respiratory function test data performed during the preoperative check-up
* Subject in exclusion period required by another protocol
* Pregnant or lactating woman, patient unable to give consent, protected adult, vulnerable persons (according to French Health Code articles L.1121-6, L.1121-7, L.1211-8, L.1211-9)
* Subject deprived of liberty by judicial or administrative decision
* Participation of the subject in another interventional protocol
* Failure to properly inform the patient (e.g. a language barrier)

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-12-16 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in: Oxygen pulse (mL O2 / heart beat) | post-op (expected maximum of 4 years) versus pre-op (approximately month -1 up to day 0))
  Recorded during incremental exercise testing.

SECONDARY OUTCOMES:
Change in: Body mass index (kg/m^2) | post-op (expected maximum of 4 years) versus pre-op (approximately month -1 up to day 0))
Change in: The presence/absence of dyspnea during exercise | post-op (expected maximum of 4 years) versus pre-op (approximately month -1 up to day 0))
Change in: The presence/absence of palpitations | post-op (expected maximum of 4 years) versus pre-op (approximately month -1 up to day 0))
Change in: The presence/absence of psychosocial impact | post-op (expected maximum of 4 years) versus pre-op (approximately month -1 up to day 0))
Change in: VO2MAX (ml/kg/min) | post-op (expected maximum of 4 years) versus pre-op (approximately month -1 up to day 0))
  Maximum oxygen consumption during incremental exercise testing.
Change in: VO2MAX (% predicted) | post-op (expected maximum of 4 years) versus pre-op (approximately month -1 up to day 0))
  Maximum oxygen consumption during incremental exercise testing.
Change in: Maximum heart rate (bpm) | post-op (expected maximum of 4 years) versus pre-op (approximately month -1 up to day 0))
  Maximum heart rate during incremental exercise testing.
Change in: Presence/absence of an anomaly in oxygen pulse | post-op (expected maximum of 4 years) versus pre-op (approximately month -1 up to day 0))
  Presence/absence of an anomaly in oxygen pulse during incremental exercise testing.
Change in: Ventilatory threshold (% of VO2MAX) | post-op (expected maximum of 4 years) versus pre-op (approximately month -1 up to day 0))
  The ventilatory threshold during incremental exercise testing.
Change in: Breathing Reserve (% of maximum voluntary ventilation) | post-op (expected maximum of 4 years) versus pre-op (approximately month -1 up to day 0))
  The breathing reserved during incremental exercise testing.
Change in: Forced expiratory volume in 1 second (liters) | post-op (expected maximum of 4 years) versus pre-op (approximately month -1 up to day 0))
Change in: Forced expiratory volume in 1 second (% predicted) | post-op (expected maximum of 4 years) versus pre-op (approximately month -1 up to day 0))
Change in: Forced vital capacity (liters) | post-op (expected maximum of 4 years) versus pre-op (approximately month -1 up to day 0))
Change in: Forced vital capacity (% predicted) | post-op (expected maximum of 4 years) versus pre-op (approximately month -1 up to day 0))
Change in: Forced expiratory volume in 1 second (litres) / forced vital capacity (litres) | post-op (expected maximum of 4 years) versus pre-op (approximately month -1 up to day 0))
Change in: Residual volume (liters) | post-op (expected maximum of 4 years) versus pre-op (approximately month -1 up to day 0))
Change in: Residual volume (% predicted) | post-op (expected maximum of 4 years) versus pre-op (approximately month -1 up to day 0))
Change in: Total lung capacity (liters) | post-op (expected maximum of 4 years) versus pre-op (approximately month -1 up to day 0))
Change in: Total lung capacity (% predicted) | post-op (expected maximum of 4 years) versus pre-op (approximately month -1 up to day 0))
Change in: Residual volume / Total lung capacity (liters/liters) | post-op (expected maximum of 4 years) versus pre-op (approximately month -1 up to day 0))
Change in: Functional residual capacity (liters) | post-op (expected maximum of 4 years) versus pre-op (approximately month -1 up to day 0))
Change in: Functional residual capacity (% predicted) | post-op (expected maximum of 4 years) versus pre-op (approximately month -1 up to day 0))
The SF36 questionnaire | post-op (expected maximum of 4 years)
  This is a general health related quality of life questionnaire.
The Body Esteem Scale | post-op (expected maximum of 4 years)
  This questionnaire treats body esteem.
The Rosenberg Self Esteem Scale | post-op (expected maximum of 4 years)
  This questionnaire treats self esteem.
Complications | per-op up to expected maximum of 4 years
Blood pressure (average, mmHg) | during surgery (day 0)
  Per-operative hemodynamic measures
Pulse | during surgery (day 0)
  Per-operative hemodynamic measures
Oxygen saturation (SpO2, %) | during surgery (day 0)
  Per-operative hemodynamic measures
Cardiac index (liters/min/m^2) | during surgery (day 0)
  Per-operative hemodynamic measures
Variation in ejection volume (%) | during surgery (day 0)
  Per-operative hemodynamic measures
Indexed systolic ejection volume (ml/beat/m2) | during surgery (day 0)
  Per-operative hemodynamic measures
Cumulative dose of vasopressors | during surgery (day 0)
  Per-operative hemodynamic measures

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Solovei, MD, Principal Investigator — University Hospitals of Montpellier, France
Locations (1):
- Hôpital Arnaud de Villeneuve - CHU de Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Suehs CM, Molinari N, Bourdin A, Solovei L. Change in cardiorespiratory parameters following surgical correction of pectus excavatum: protocol for the historical-prospective HeartSoar cohort. BMJ Open. 2023 Jun 15;13(6):e070891. doi: 10.1136/bmjopen-2022-070891. PMID 37321811